CLINICAL TRIAL: NCT01259882
Title: A Double Blind (3rd Party Open) Randomized, Placebo Controlled, Crossover Dose Escalation Study To Investigate The Safety, Toleration, Pharmacokinetics And Exploratory Pharmacodynamics Of PF-05089771 In Healthy Volunteers
Brief Title: A Single Dose Escalation Study In Healthy Volunteers To Determine The Pharmacokinetics, Safety And Tolerability Of PF-05089771 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B3291001
Record Dates: First submitted 2010-11-30; First posted 2010-12-14 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Pain
Keywords: Pharmacokinetics Safety Tolerability Pharmacodynamics
MeSH Terms: conditions — Pain | interventions — PF-05089771

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1: Experimental intervention: PF-05089771 or placebo (Experimental): Cohort 1
  Interventions: Drug: PF-05089771
- Cohort 2: Experimental intervention: PF-05089771 or placebo (Experimental): Cohort 2
  Interventions: Drug: PF-05089771
- Cohort 3: Experimental intervention: PF-05089771 or placebo (Experimental): Cohort 3
  Interventions: Drug: PF-05089771
- Cohort 4: Experimental intervention: PF-05089771 or placebo (Experimental): Cohort 4
  Interventions: Drug: PF-05089771
- Cohort 5: Experimental intervention: PF-05089771 or placebo (Experimental): Cohort 5
  Interventions: Drug: PF-05089771
- Cohort 6: Experimental intervention: PF-05089771 or placebo (Experimental): Cohort 6
  Interventions: Drug: PF-05089771

INTERVENTIONS:
Drug: PF-05089771 — Subjects will receive single ascending doses of PF-05089771 or placebo to investigate the safety/tolerability and PK of PF-05089771. The PK of alternative formulations of PF-05089771 and the effect of food on PK may also be investigated.
  Arms: Cohort 1: Experimental intervention: PF-05089771 or placebo
Drug: PF-05089771 — Subjects will receive single ascending doses of PF-05089771 or placebo to investigate the safety/tolerability and PK of PF-05089771. The PK of alternative formulations of PF-05089771 and the effect of food on PK may also be investigated.
  Arms: Cohort 2: Experimental intervention: PF-05089771 or placebo
Drug: PF-05089771 — Subjects will receive single doses of PF-05089771 or placebo in a fully randomized crossover design. The investigation of the safety/tolerability and PK of PF-05089771 will occur. In addition the exploratory pharmacodynamics of PF-05089771 will be investigated using novel biomarkers.
  Arms: Cohort 3: Experimental intervention: PF-05089771 or placebo
Drug: PF-05089771 — Subjects will receive single doses of PF-05089771 or placebo in a fully randomized crossover design. The investigation of the safety/tolerability and PK of PF-05089771 will occur.
  Arms: Cohort 4: Experimental intervention: PF-05089771 or placebo
Drug: PF-05089771 — Subjects will receive single doses of PF-05089771 or placebo in a fully randomized crossover design. The investigation of the safety/tolerability and PK of PF-05089771 will occur.
  Arms: Cohort 5: Experimental intervention: PF-05089771 or placebo
Drug: PF-05089771 — Subjects will receive single doses of PF-05089771 or placebo in a fully randomized crossover design. The investigation of the safety/tolerability and PK of PF-05089771 will occur.
  Arms: Cohort 6: Experimental intervention: PF-05089771 or placebo

SUMMARY:
This is a two part study. The purpose of the first part is primarily to determine the safety and toleration and pharmacokinetics of PF-05089771 following single escalating doses. Secondary objectives will be to investigate the PK of an alternative formulation of PF-05089771 and the effect of food on the PK of PF-05089771. The second part of the study will focus on investigation of the exploratory pharmacodynamics of PF-05089771 using novel biomarkers in healthy volunteers. The doses selected in Part B will have been administered previously in Part A of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects or female subjects of non-child bearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (e.g., gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 21 drinks/week (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug within 60 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* 12-lead ECG demonstrating QTc >450 msec at screening. If QTc exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* Females of child bearing potential.
* Use of prescription or non-prescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements must be discontinued 28 days prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of 1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing. History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of PF-05089771. | Days 1-3
Maximum concentration (Cmax) for PF-05089771 in plasma (measured in ng/mL) | Days 1-3
Tmax = Time of maximum concentration of PF-05089771 in plasma (hr) | Days 1-3
AUClast = Area under the curve from the time of dosing to the last data point taken (ng.hr/mL) | Days 1-3
MRT = Mean residence time of PF-05089771 in the body (hr) | Days 1-3

SECONDARY OUTCOMES:
Heat Pain Perception Threshold (HPPT). Measured by applying a heat thermode to the thigh for 1 minute at 47oC. HPPT will be measured at 3 separate doses plus placebo in 12 healthy volunteers. | Hours 1-6 post dose.
Long Thermal Stimulation (LTS). Measured by applying a heat thermode to the thigh at 48oC for 5 seconds. will be measured at 3 separate doses plus placebo in 12 healthy volunteers | Hours 1-6 post dose.
Odor threshold (Sniffin' Sticks). Measured with Sniffin Sticks. Will be measured at 3 separate doses plus placebo in 12 healthy volunteers | Hours 1-6 post dose.
Urine: Aet (amount excreted in urine), Aet% and CLr for selected doses dependent on the emerging pharmacokinetics of PF-05089771 where t = 24 hours. | Up to 24 hours
AUCinf = Area under the curve from the time of dosing extrapolated to infinity (ng.hr/mL) | Days 1-3
AUC24 = Area under the curve from the time of dosing to 24 hours post dose (ng.hr/mL) | Days 1-3
CI/F = Clearance of PF-05089771 from plasma corrected for systemic compound availability (L/hr) | Days 1-3
t½ = Elimination half life of PF-05089771 (hr) | Days 1-3
C8 hour = concentration of PF-05089771 in the plasma 8 hours post dose (ng/mL) | Days 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3291001&StudyName=A%20Single%20Dose%20Escalation%20Study%20In%20Healthy%20Volunteers%20To%20Determine%20The%20Pharmacokinetics%2C%20Safety%20And%20Tolerability%20Of%20PF-05089771%20In%20Health